CLINICAL TRIAL: NCT05725941
Title: The Effectiveness of Spiral Strapping on Upper Limb Functions in Individuals with Stroke
Brief Title: Spiral Strapping for Improving Upper Limb Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Collaborators: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Abd El Kafy, Professor of Physical Therapy, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RI-4-0588
Record Dates: First submitted 2023-01-23; First posted 2023-02-13 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2023-01

CONDITIONS: Stroke; Splints; Physical Disability
Keywords: Stroke; Upper Limb Functions; Spiral Strapping
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Individuals who will participate in the control group will receive a traditional functional exercise training protocol (conventional physiotherapy program) for one hour. It will focus on the enhancement of muscle strength, joint range of motion, arm &hand activities, and daily living functions of the affected upper limbs.
  The treatment, for the control group, will be conducted over a period of 4 successive weeks, with 3 sessions per week.
  Interventions: Other: Traditional upper limb functional exercise training
- Experimental Group (Experimental): Participants in the experimental group will receive the conventional treatment program similar to that will be provided to the control group. The treatment, for the experimental group, will be conducted over a period of 4 successive weeks, with 3 sessions per week.
  Moreover, they will ¬wear an upper limb spiral strapping system with a hand splint 8 hours daily/ 6 days per week.
  Interventions: Device: TogRite stretch Strapping; Other: Traditional upper limb functional exercise training

INTERVENTIONS:
Device: TogRite stretch Strapping — it is a machine washable and highly durable elastic strap that maintains its recoil strength for a long-lasting period. It is made of latex-free materials. The TogRite Strapping can be used to support the weakened parts of the body and adjust or modify the position and posture of different body parts.
  Arms: Experimental Group
Other: Traditional upper limb functional exercise training — The traditional upper limb functional exercise training will focus on the enhancement of muscle strength, joint range of motion, arm &hand activities, and daily living functions of the affected upper limbs.

SUMMARY:
Upper limb recovery after stroke is unacceptably poor with almost half of stroke survivors likely to regain some functional use. The rehabilitation process for upper extremity for individuals with stroke is of long duration and clinicians face the challenge of identifying a variety of assistive appliances that may be adapted and graded to facilitate this process. One of these appliances that is widely used in rehabilitation is splint and strapping. Therefore, this study aims to investigate the effectiveness of this modality in rehabilitation of the upper limb in stroke survivors.

DETAILED DESCRIPTION:
Stroke often results in spasticity and associated motor impairments in the upper limb Spasticity in the upper limb commonly interferes with its motor activities, and results in impairments in the upper limb muscles. Persistent upper limb impairments can lead to limitations in activities of daily living, and quality of life. Assistive devices to facilitate the use of the hemiplegic upper extremity are considered to be the most important modalities in improving the functions of the upper limb. The splint is one of the most assistive tools in the rehabilitation of such individuals. The supportive and corrective functions provided by upper limb and hand splints have been shown to inhibit spasticity and promote the capabilities of the upper limb in individuals with stroke This study aims to evaluate the effectiveness of spiral strapping on inhibition of spasticity and improving upper limb functions in individuals with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were as follow:

* Participants were diagnosed as chronic stroke patients.
* Participants were selected to be in the spastic phase.
* The degree of spasticity in the affected upper limbs, was ranged between grades (1, 1+&2) according to Modified Ashworth Scale.
* Participants were all between 50 and 60 years old, of both sexes.
* Participants were cognitively able to understand and follow instructions.
* Participants had the ability to extend their wrist joints at least 20° and ﬁngers 10° from full ﬂexion. This range allowed participants to engage easily in performing a designed functional program.

Exclusion Criteria:

The exclusion criteria were as follow:

* Participants who were with any orthopedic condition or fixed deformity that interfere with the upper limb functions.
* Participants who were with spasticity of more than score 2 according to the Modified Ashworth Scale.
* Participants who had cognitive or perceptual problems.
* Participants with seizures, visual impairments, or auditory problems.
* Participants who had shoulder pain on a visual analogue scale of > 6/10.
* Participants who had Botulinum Toxin in the upper extremity musculature six months before baseline assessment.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in the score of The Action Research Arm Test (test that assess the change in upper extremity functions) | [Data was collected at baseline, and 4weeks after intervention commencement.] (i.e. Difference between The Action Research Arm Test Score at both baseline and completion of 4 weeks of intervention)
  The Action Research Arm Test (ARAT) is an evaluative measure to assess specific changes in limb function among individuals with hemiplegia. It assesses a patient's ability to handle objects differing in size, weight and shape and therefore can be considered to be an arm-specific measure of activity limitation. The ARAT consists of 19 items grouped into four subscales: grasp, grip, pinch, and gross movement. The ARAT is scored on a four-level ordinal scale (0-3): 0 = cannot perform any part of the test, 1 = performs partially, 2 = take long time to complete the test, and 3 = performs the test normally. The total score on the ARAT ranges from 0 to 57, with the lowest score indicating that no movements can be performed, and the upper score indicating normal performance. Thus, the higher the score a patient get after completion of the treatment program compared to the baseline score, the better the improvement in upper extremity motor functions.
Change in the Modified Ashworth Scale (scale that assess the change in muscle tone) | [Data was collected at baseline, and 4weeks after intervention commencement.] (i.e. Difference between The Action Research Arm Test Score at both baseline and completion of 4 weeks of intervention)
  Modified Ashworth Scale was used to evaluate the degree of spasticity in the involved upper limb in the elbow and wrist joints. MAS is a valid and a reliable scale to evaluate the degree of muscle tone for all participants pre and post treatment. It is scored on a 6 -graded ordinal scale.
Change in the upper limb' joints range of motion (in degree) | [Data was collected at baseline, and 4 weeks after intervention commencement.] (i.e. Difference between The Action Research Arm Test Score at both baseline and completion of 4 weeks of intervention)
  Digital Goniometer was used to evaluate the following joints range of motion (shoulder abduction& external rotation, elbow extension and forearm supination). The Digital Goniometer has used a sensor to calculate the amount of joint range of motion in degrees to measure the true range of motion value.

SECONDARY OUTCOMES:
Change in the Hand Grip Strength of the involved upper extremity (Kg) (which indicate the change of the strength of the involved hand muscles in patients with stroke). | [Data was collected at baseline, and 4 weeks after intervention commencement.] (i.e. Difference between The Action Research Arm Test Score at both baseline and completion of 4 weeks of intervention)
  Hand Grip Dynamometer was used to assess the change in the strength of the hand muscles of the involved upper extremity. The higher the score of the hand grip after completion of the treatment program compared to the baseline score, the better the improvement of hand functional abilities.

CONTACTS AND LOCATIONS:
Locations (1):
- Ehab Mohamed Abd El Kafy, Mecca, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
- The data available is Case-by-case basis at the discretion of the Primary Sponsor
Supporting Information: SAP
Time Frame: Start Date: Beginning one year following main results publication End Date: Ending two years following main results publication
Access Criteria: Data can be obtained by the Principal Investigator. Email Address: emkafy@uqu.edu.sa